CLINICAL TRIAL: NCT04423367
Title: Safety and Efficacy of Bortezomib Plus Dexamethasone for Acquired Pure Red Cell Aplasia Failure or Relapse After First-line Treatment: A Prospective Phase II Trial
Brief Title: Bortezomib Plus Dexamethasone for Acquired Pure Red Cell Aplasia Failure or Relapse After First-line Treatment
Acronym: BID-PERAL
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT2020010
Record Dates: First submitted 2020-06-05; First posted 2020-06-09 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2024-11

CONDITIONS: Acquired Pure Red Cell Aplasia
Keywords: Acquired Pure Red Cell Aplasia; PRCA; Failure or Relapse after First-line Treatment
MeSH Terms: interventions — Bortezomib; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- bortezomib/dexamethasone (Experimental): Enrolled patients will receive the combination therapy of bortezomib and dexamethasone.
  Interventions: Drug: bortezomib/dexamethasone

INTERVENTIONS:
Drug: bortezomib/dexamethasone — Enrolled patients would receive the combination therapy of bortezomib and dexamethasone.

SUMMARY:
This is an open-label, single-arm study to evaluate the safety and efficacy of bortezomib plus dexamethasone for acquired pure red cell aplasia failure or relapse after first-line treatment.

ELIGIBILITY:
Inclusion Criteria:

* ECOG ≤ 2.
* Age from 18 to 70.
* Diagnosed with acquired pure red cell aplasia.
* Meets the criteria of first-line treatment failure or relapse.
* Organs in good function.
* Signed informed consent.

Exclusion Criteria:

* Nursing woman.
* Active bacterial, virus, fungal or parasitic infection, including HIV infection, HBsAg or HBV DNA positive, HCV DNA positive, etc.
* Secondary PRCA caused by lymphoproliferative disorders, including large granular lymphocytic leukemia, waldenström macroglobulinemia, small lymphocytic lymphoma/chronic lymphocytic leukemia, etc.
* Secondary PRCA caused by either smoldering multiple myeloma or symptomatic multiple myeloma.
* Secondary PRCA caused by either ABO major mismatched stem cell transplantation or organ transplantation.
* Secondary PRCA caused by solid tumors except for thymoma.
* Secondary PRCA caused by drugs or pregnancy.
* Secondary PRCA caused by the B19 virus.
* Have contraindications for glucocorticoids, or unable to tolerate glucocorticoids for comorbidities.
* Previously received treatment in other trials within 4 weeks before enrollment.
* Previously treated with the proteasome inhibitor.
* Experience active hemorrhage condition, including gastrointestinal bleeding, respiratory tract bleeding and central nervous system bleeding within 2 months before enrollment or during bortezomib/dexamethasone treatment.
* Have a history of malignant tumors.
* Have a history of mental illness.
* Inability to understand or to follow study procedures.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2020-09-13 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
Overall response rate | within 12 weeks

SECONDARY OUTCOMES:
Frequency and severity of adverse events and severe adverse events | within 12 weeks
Relapse free survival | within 24 and 48 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jun Shi, PhD, Principal Investigator — Institute of Hematology & Blood Diseases Hospital, China
Locations (3):
- China (3):
  - Zhoukou Central Hospital, Zhoukou, Henan
  - The Second Affilated Hospital of Shandong First Medical University, Tai’an, Shandong
  - Regenerative Medicine Center, Tianjin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zhang L, Chen N, Xu Z, Liang Q, Pan H, Zhao J, Fang L, Shi J. Good treatment-free survival of monoclonal gammopathy of undetermined significance associated pure red cell aplasia after bortezomib plus dexamethasone. Blood Cells Mol Dis. 2021 Jul;89:102573. doi: 10.1016/j.bcmd.2021.102573. Epub 2021 Apr 27. PMID 33957358